CLINICAL TRIAL: NCT02918760
Title: Oral Gabapentin in Management of Chronic Pelvic Pain in Females: A Randomised Placebo-controlled Study.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ahmed Elnaggar, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIN-02-01-2016
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Pelvic Pain
Keywords: Gabapentin, chronic pelvic pain.
MeSH Terms: conditions — Pelvic Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): This group will include (32) women according to inclusion and exclusion criteria and will receive a card of Gabapentin which will be taken orally by the patient at home three times daily and maximum dose 2700mg per day by 300 mg increments each week until sufficient pain relief, or the occurrence of side effects such as dizziness, somnolence, edema and ataxia.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Group B (controls):This group will include (32) women according to inclusion and exclusion criteria and will receive a card of placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — This group will include (32) women according to inclusion and exclusion criteria and will receive a card of Gabapentin which will be taken orally by the patient at home three times daily and maximum dose 2700mg per day by 300 mg increments each week until sufficient pain relief, or the occurrence of side effects such as dizziness, somnolence, edema and ataxia.
  Arms: Gabapentin
Other: Placebo — Group B (controls):This group will include (32) women according to inclusion and exclusion criteria and will receive a card of placebo.
  Arms: Placebo

SUMMARY:
Aim :The aim of this study is to evaluate the efficacy of oral Gabapentin in the treatment of chronic pelvic pain in females.

The study is designed as a randomised, placebo-controlled, clinical trial.32 patients will be enrolled each arm.

Group A (cases):

This group will include (32) women according to inclusion and exclusion criteria and will receive a card of Gabapentin which will be taken orally by the patient at home three times daily and maximum dose 2700mg per day by 300 mg increments each week until sufficient pain relief, or the occurrence of side effects such as dizziness, somnolence, edema and ataxia. Group B (controls):This group will include (32) women .

Assessment of the patient's pain during the physical examination will be done using the Visual Analogue Scale (VAS). The patient will be asked to place a mark on a drawn 10 cm line at a point which is corresponding to the intensity of her pain. One end of the line denotes no pain and the other end of the line indicates that pain is as bad as it can be (the worst pain).the distance in cm from the low end of VAS to the patient's mark will be used (it gives a number.Questionnaire: will be given to all participants at randomization (0 months) , at 3 months and at 6 months to assess the degree of pain improvement via VAS.

Patients' overall satisfaction with their pain treatment &Side effect recording (e.g., dizziness, somnolence, mood changes, appetite and poor concentration).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe chronic pelvic pain for at least 6 months.
* Pain was unrelated exclusively to menstruation.
* Pain incompletely relieved by Non-steroidal Ant-inflammatory drugs.
* Patients had regular menstrual cycles for 3 months.
* Patient receiving regular, effective contraceptive method.

Exclusion Criteria:

* Pregnancy or planning of pregnancy in next 6 months.
* Breast feeding.
* Acute pelvic infection.
* Known history of hypersensitivity to Gabapentin.
* Patients with severe renal or hepatic failure.
* Women with previous diagnosis of endometriosis confirmed by laparoscopy.
* Women with previous diagnosis of Malignancy.
* Plans for surgery in next 6 months.
* Women with chronic or recurrent gastrointestinal disease, including irritable bowel syndrome.
* Women with histories of alcohol use or other chronic tranquilizers. Patients refuse to sign an informed consent form.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain score improvement | 6 months

SECONDARY OUTCOMES:
Side effect recording | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel hafeez, A.professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] AbdelHafeez MA, Reda A, Elnaggar A, El-Zeneiny H, Mokhles JM. Gabapentin for the management of chronic pelvic pain in women. Arch Gynecol Obstet. 2019 Nov;300(5):1271-1277. doi: 10.1007/s00404-019-05272-z. Epub 2019 Aug 21. PMID 31435774